CLINICAL TRIAL: NCT05064579
Title: Towards an Algorithmic Approach to Asthma Management: Collaborative Definition of Algorithm Objectives With Families
Acronym: COPA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210819; 2021-A00041-40 (Other: ID RCB number)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Childhood Asthma
Keywords: Childhood asthma; Algorithms for managing childhood asthma; Big data; Artificial intelligence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with asthma: Children and adolescents aged 8 to 17 years old with a doctor's diagnosis of asthma and controller asthma treatment
  Interventions: Other: Questionnaires
- Holders of parental authority: Holders of parental authority of patients with asthma described in group A
  Interventions: Other: Questionnaires
- Doctors: Doctors caring for patients with asthma described in group A
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaire in two parts: one part on the objectives related to taking the treatment and the objectives related to the treatment modality and a second part on the general characteristics of each participant and the characteristics of the child's asthma.

SUMMARY:
Using "big data" and artificial intelligence techniques, it becomes possible to envision algorithms for managing childhood asthma on a daily basis.

In order to develop such tools, it is necessary to determine with asthma stakeholders (children, parents, doctors) the parameters that future algorithms should seek to maximize / minimize.

The main objective of the study is to quantify the respective importance of each of the goals that children with asthma, parents, and their doctors seek to achieve when taking / supervising / prescribing a background therapy.

DETAILED DESCRIPTION:
Using "big data" and artificial intelligence techniques, it becomes possible to envision algorithms for managing childhood asthma on a daily basis.

In order to develop such tools, it is necessary to determine with asthma stakeholders (children, parents, doctors) the parameters that future algorithms should seek to maximize / minimize.

The main objective of the study is to quantify the respective importance of each of the goals that children with asthma, parents, and their doctors seek to achieve when taking / supervising / prescribing a background therapy.

To do this, parents and children fill out a paper questionnaire, which is completed by their doctor, when they come to the hospital for consultation, hospitalization, or to perform lung function tests.

Concerning children and parents, these questionnaires include a part aimed at prioritizing each person's objectives and a second part collecting general information regarding their characteristics (age, sex, asthma history, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Minor patients aged 8 years to 17 years and 11 months inclusive with a diagnosis of asthma made by a doctor and a basic treatment for asthma
* Holders of parental authority for patients meeting the above criteria
* Doctors caring for children with asthma
* Information and non-opposition of holders of parental authority and minor patients to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Difficulties in French writing and / or speaking

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited in hospitals in the Ile-de-france region
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Mean score attributed to each goal | Day 0
  Children, their parents (or holders of parental authority), and their doctors will be asked to allocate 20 points to 7 goals they want to prevent with the asthma controller treatment, and another 20 points to 5 goals regarding their treatment modality (more discreet, easier to take, etc). The score for each goal will range from 0 (objective not important to the respondent) to 20 (objective of major importance to the respondent).

SECONDARY OUTCOMES:
Correlation of goals between respondents | Day 0
  For each goal, the correlation of the scores attributed by children, their parents, and their doctors, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: David Drummond, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Louis Mourier, Colombes
  - Hôpital Trousseau-Allergologie pédiatrique, Paris
  - Hôpital Trousseau-Pneumologie pédiatrique, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masrour O, Personnic J, Amat F, Abou Taam R, Prevost B, Lezmi G, Gonsard A, Nathan N, Pirojoc A, Delacourt C, Wanin S, Drummond D. Objectives for algorithmic decision-making systems in childhood asthma: Perspectives of children, parents, and physicians. Digit Health. 2024 Feb 21;10:20552076241227285. doi: 10.1177/20552076241227285. eCollection 2024 Jan-Dec. PMID 38389509